CLINICAL TRIAL: NCT02453269
Title: Outcome of a 1-year Transdisciplinary Program Against Childhood Obesity
Brief Title: Transdisciplinary Program Against Childhood Obesity
Acronym: OTPACO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fortaleza University (Other)
Responsible Party: Principal Investigator, Carminda Maria Goersch Fontenele Lamboglia, Outcome of a 1-year transdisciplinary program against childhood obesity, Fortaleza University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRANS 123
Record Dates: First submitted 2015-04-13; First posted 2015-05-25 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Childhood Obesity
Keywords: Obesity; Children; Health Colective
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transdisciplinary program (Experimental): Children in G1 were submitted to a transdisciplinary intervention once a week. Each child received a nutritional education kit including four games ("Cool Diet", a board game, a memory game and a word search puzzle) and an interactive booklet containing).
  Interventions: Behavioral: Transdisciplinary program
- Control group (No Intervention): The children in the control group (G2) were not exposed to interventions.

INTERVENTIONS:
Behavioral: Transdisciplinary program
  Arms: Transdisciplinary program

SUMMARY:
The purpose of this study was to evaluate the outcome of a 1-year transdisciplinary program against childhood obesity.

DETAILED DESCRIPTION:
The study was quasi-experimental with a quantitative approach.5 Epidemiologically, the study may be characterized as a controlled, randomized trial. Twenty participants were selected non-randomly from an elementary school in Fortaleza, Brazil. The parents or caretakers of the participants gave their informed written consent. The 20 participants were distributed randomly into two groups, G1 (intervention, n=10) and G2 (control, n=10). Six children did not complete the study protocol: three in G1 due to insufficient attendance, and three in G2 for unspecified reasons. To be eligible for the study, children should i) be overweight or obese in accordance with the definition given above6, ii) be considered healthy by a physician after undergoing a clinical examination, iii) attend the transdisciplinary intervention sessions once a week (minimum attendance required: 90%) and iv) be authorized to participate by their parents or caretakers. The children in the control group were not submitted to the intervention and were not participating in any other program involving obesity control or supervised physical activity. All children (G1+G2) were instructed to maintain their habitual level of physical activity and attend the school's regular physical education classes. The latter were scheduled twice a month during the first term and four times a month during the second. The decision to increase the frequency was made by the school's director in acknowledgment of the importance of physical activity, but the change affected the two groups equally. Children were ineligible if they had chronic diseases (defined as diseases requiring continuous therapy), mental disorders or cognitive impairments which might interfere with communication, or used a pacemaker, or declined participation. Children in G1 missing more than 10% of the total intervention sessions were excluded from the sample. The study was conducted at an elementary school in Fortaleza, Brazil, maintained by the Edson Queiroz Foundation/UNIFOR. Data were collected at baseline in May 2013 (pre-test) and after one year of intervention, in May 2014 (post-test), as part of the transdisciplinary program against childhood obesity. Children in G1 were submitted to a transdisciplinary intervention once a week. Each child received a nutritional education kit including four games ("Cool Diet", a board game, a memory game and a word search puzzle) and an interactive booklet containing illustrations of foods selected from the participants' cultural context (Northeastern Brazil). The kit was validated by Munguba. The children in the control group (G2) were not exposed to interventions during the study period. They attended the school's regular physical education classes, but were excluded from the sample if they joined any other physical activity or weight control program. At the end of the study, the children in G2 received the booklet described above, including the results of the physical fitness evaluation. Talks about the importance of physical activity and healthy food in this group were scheduled for early 2015. Upon the first visit, all participants were given a physical evaluation (BMI, height and waist circumference) following the procedures standardized by Lohman, Roche and Martorell. The body composition was determined by bioelectrical impedance (Bodystat 1500 MMD) upon the second visit. Upon the first, the children were instructed in how to prepare for the test: abstain from food and drink (4 hours before), exercise (12 hours before), alcohol (24 hours before) and diuretic medication (7 days before), and urinate 30 min before the test. The subject is measured lying down, with electrodes attached to hands and feet. The muscular fitness assessment was based on FitnessGram®, a criterion-referenced test, but was limited to flexibility and abdominal muscle strength/endurance. The evaluation of sexual maturity was based on the age at menarche in girls and on armpit hair development in boys. The purpose of this evaluation was to identify each participant's stage of growth, development and maturity.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for the study, children should

  * be overweight or obese in accordance with the definition given above6,
  * be considered healthy by a physician after undergoing a clinical examination,
  * attend the transdisciplinary intervention sessions once a week (minimum attendance required: 90%)
  * be authorized to participate by their parents or caretakers.
* The children in the control group were not submitted to the intervention and were not participating in any other program involving obesity control or supervised physical activity.
* All children (G1+G2) were instructed to maintain their habitual level of physical activity and attend the school's regular physical education classes.
* The latter were scheduled twice a month during the first term and four times a month during the second.
* The decision to increase the frequency was made by the school's director in acknowledgment of the importance of physical activity, but the change affected the two groups equally.

Exclusion Criteria:

* Children were ineligible if they had chronic diseases (defined as diseases requiring continuous therapy), mental disorders or cognitive impairments which might interfere with communication, or used a pacemaker, or declined participation.
* Children in G1 missing more than 10% of the total intervention sessions were excluded from the sample.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Height (cm) (outcome) | Participants were followed for the duration of one year
Body mass (kg) (outcome) | Participants were followed for the duration of one year
Body mass index (kg/m2) (outcome) | Participants were followed for the duration of one year
Waist circumference (cm) (outcome) | Participants were followed for the duration of one year
Waist circunference/height ratio (outcome) | Participants were followed for the duration of one year
Body fat percentage (%) (outcome) | Participants were followed for the duration of one year
Fat body mass (kg) (outcome) | Participants were followed for the duration of one year
Lean body mass (kg) (outcome) | Participants were followed for the duration of one year
Abdominal strength (repetition) (outcome) | Participants were followed for the duration of one year
Flexibility (cm) (outcome) | Participants were followed for the duration of one year

CONTACTS AND LOCATIONS:
Locations (1):
- Carminda Maria Goersch Fontenele Lamboglia, Fortaleza, Ceará, Brazil